CLINICAL TRIAL: NCT04177472
Title: MAGIC: a Family Based Feeding Intervention Program
Brief Title: Mothers and CareGivers Investing in Children
Acronym: MAGIC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: St. David's Foundation (Unknown); National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry); Egg Nutrition Center (Other); National Pork Board (Other)
Responsible Party: Principal Investigator, Deborah Jacobvitz, Phyllis L. Richards Endowed Professor in Child Development, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UT Austin IRB#2015040017
Record Dates: First submitted 2019-10-25; First posted 2019-11-26 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Obesity, Childhood; Parenting
Keywords: nutrition; parenting; intergenerational feeding influences; sensitive feeding
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Primary - BMI percentile at 12 months of age, and 24 months of age
  Secondary- Proportion of infants with BMI percentile >85th at 12 months of age, and 24 months of age
  Anthropometrics measured directly by trained study staff
  Infant dietary intake of fruits and vegetables, animal source foods, whole grains, desserts and sweets, and salty snacks at 10 to 11 months.
  Measured at 10 months using an Infant Diet History questionnaire adapted from the Infant Feeding Practices Study II. Measured at 10 months using the Nutrition Data System for Research (NDSR)
  Responsive feeding measured using the Infant Feeding Styles Questionnaire (IFSQ) full scale and Chatoor's feeding scale at 10 to 11 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Obesity Prevention Group (Experimental): Parents will be provided with responsive feeding coaching to help them recognize hunger and satiety cues and nutrition coaching that involves recommending a sequence of introducing complementary foods that corresponds with food textures and feeding styles, breast/bottle weaning, healthy snacking and hands on demonstrations for healthy food options.
  Interventions: Behavioral: Obesity Prevention Group
- Infant Safety and Injury Prevention Group (Active Comparator): Parents will be provided with information about safe sleeping, car seats, baby-proofing, etc., delivered during virtual visits, participant binder and newsletter.
  Interventions: Behavioral: Infant Safety and Injury Prevention Group
- Obesity Prevention Group + Food Boxes (Experimental): Parents will be provided with responsive feeding coaching to help them recognize hunger and satiety cues and nutrition coaching that involves recommending a sequence of introducing complementary foods that corresponds with food textures and feeding styles, breast/bottle weaning, healthy snacking and hands on demonstrations for healthy food options. Parents will also be provided with grocery items (fruits, vegetables, meat) prior to each intervention visit to facilitate a healthy family diet.
  Interventions: Behavioral: Obesity Prevention Group + Food Boxes

INTERVENTIONS:
Behavioral: Obesity Prevention Group — Parents will be provided with responsive feeding coaching to help them recognize hunger and satiety cues and nutrition coaching that involves recommending a sequence of introducing complementary foods that corresponds with food textures and feeding styles, breast/bottle weaning, healthy snacking and hands on demonstrations for healthy food options.
  Arms: Obesity Prevention Group
Behavioral: Obesity Prevention Group + Food Boxes — Parents will be provided with responsive feeding coaching to help them recognize hunger and satiety cues and nutrition coaching that involves recommending a sequence of introducing complementary foods that corresponds with food textures and feeding styles, breast/bottle weaning, healthy snacking and hands on demonstrations for healthy food options. Parents will also be provided with grocery items (fruits, vegetables, meat) prior to each intervention visit to facilitate a healthy family diet.
  Arms: Obesity Prevention Group + Food Boxes
Behavioral: Infant Safety and Injury Prevention Group — Parents will be provided with information about safe sleeping, car seats, baby-proofing, etc., delivered during home visits, newsletters, and reinforcing text messages.
  Arms: Infant Safety and Injury Prevention Group

SUMMARY:
The incidence of childhood obesity in the United States has steadily increased over the past 30 years but has begun to level off in recent years. Epidemiological evidence indicates that obesity may transmitted across multiple generations. The current study seeks to: 1) evaluate the extent to which mothers and other important caregivers affect their mothers' parenting; 2) examine whether an intervention aimed at improving diet quality and enhancing responsive feeding to improves parental responsivity and feeding behavior and infants' weight trajectories over time; 3) examine the effects of early life feeding and caregiver sensitivity on health and development; and 4) examine feasibility of food distribution along with the feeding intervention.

DETAILED DESCRIPTION:
The incidence of childhood obesity in the United States has steadily increased over the past 30 years, but has begun to level off in recent years. Children from minority groups may be disproportionately affected, such that Hispanic and non-Hispanic Black children have greater weight for recumbent length compared to White children. Similarly, socioeconomic status (SES) may affect child weight status. Epidemiological evidence indicates that obesity may transmitted across multiple generations. Genetics are a factor in determining weight status, but parents are largely responsible for regulating children's dietary environments. Grandparents increasingly provide care for their grandchildren, yet few studies have examined grandparent involvement or the role that grandparents or other significant caregivers play in feeding the child.

The objective of the current study is two-fold: 1) to evaluate the extent to which mothers and other caregivers affect mothers' parenting surrounding feeding their infant, beginning when the infant is first introduced to solid foods; and 2) to examine whether an intervention aimed at providing both mothers and and other important caregivers with hands-on training regarding healthy foods and responsive and sensitive feeding behaviors improves mothers' and other caregivers' responsive and sensitive behaviors and infants' weight trajectories over time. The researchers will collect both self-report data on diet, child temperament, mothers and caregiver mental health, stress and support. Observational assessments will be obtained to code co-caregiver behavior and caregiver responsiveness during feeding.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with babies aged 4 to 5 months
* Other caregivers assisting the mother with the baby.
* Babies aged 4 to 5 months

Exclusion Criteria:

* Babies with metabolic or feeding issues.
* Mothers younger than 16 years of age.

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
BMI percentile at 12 months of age | 12 months
  Anthropometrics measured by trained study staff
BMI percentile at 24 months of age | 24 months
  Anthropometrics measured by trained study staff

SECONDARY OUTCOMES:
Proportion of infants with BMI percentile >85th at 12 months of age | 12 months
  Anthropometrics measured by trained study staff
Proportion of infants with BMI percentile >85th at 24 months of age | 24 months
  Anthropometrics measured by trained study staff

OTHER OUTCOMES:
Infant dietary intake of fruits and vegetables, animal source foods, whole grains, desserts and sweets, and salty snacks at 11 months of age | 10 to 11 months of age
  Measured at 10-11 months using an Infant Diet History questionnaire adapted from the Infant Feeding Practices Study II. Measured at 10 to 11 months using the Nutrition Data System for Research (NDSR)
Responsive feeding at 10 to 11 months of age | 10 to 11 months of age
  Measured using the Infant Feeding Styles Questionnaire (IFSQ) full scale
Responsive feeding at 10 to 11 months of age | 11 months of age
  Measured during mealtime observations using the Chatoor's feeding scale.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Jacobvitz, PhD, Principal Investigator — University of Texas at Austin; Elizabeth Widen, PhD, RD, Principal Investigator — University of Texas at Austin
Locations (2):
- United States (2):
  - Sarah M. & Charles E. Seay Building, Austin, Texas
  - Dell Pediatric Research Institute, Austin, Texas

IPD SHARING:
Plan to Share IPD: No